CLINICAL TRIAL: NCT03121768
Title: A New Prognostic Model for Predicting the Outcome of Patients With Non-muscle Invasive Bladder Cancer Using Clinical Histopathological and Biological Markers
Brief Title: A New Prognostic Model for Predicting the Outcome of Patients With Non-muscle Invasive Bladder Cancer (NMIBC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abdelwahab Hashem, Msc, Mansoura University
Other Study IDs: RP/16.08.87
Record Dates: First submitted 2017-03-15; First posted 2017-04-20 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Oncology; Bladder Cancer; Superficial Bladder Cancer; Recurrence; Progression; BCG
Keywords: Prognostic Model; Bladder Cancer; Superficial Bladder Cancer; Recurrence; Progression; BCG
MeSH Terms: conditions — Neoplasms; Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Recurrence; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bladder biopsy of TURBT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective observational study to re-establish a new prognostic model for predicting the outcome in patients with non-muscle invasive bladder cancer (NMIBC) using the current recommendation regimen for intermediate and high risk groups and including all potential and highly prognostic factors.

DETAILED DESCRIPTION:
Bladder urothelial carcinoma is the most common cancer of the urinary tract and is the 7th most common cancer in males and the 7th most common cancer in females. Most of newly diagnosed cases of urothelial cancer of the bladder are non-muscle invasive (NMIBC), and including stages Ta, T1, or Carcinoma in situ (CIS). The initial management is endoscopic resection, aiming at complete removal of all visible papillary lesions, and accurate staging of the bladder tumor. The future plan is determined based on the results of histopathological diagnosis and included either re-resection or adjuvant immunotherapy.

The incidence of recurrence and progression to muscle invasive disease after resection of NMIBC reaches up to 42 % and 21%, respectively, concluding that alternative treatments are urgently required. Therefore, the development of prognostic models is of ultimate importance to minimize long-term morbidity and improve the outcome. The most commonly used stratification systems are the European Organization for Research and Treatment of Cancer (EORTC) risk tables and the The Club Urologico Espanol de Tratamiento Oncologico (CUETO) scoring model. The EORTC risk tables have been constructed based on 2596 patients diagnosed with Ta/T1 urothelial bladder carcinoma. Nevertheless, there were low number of patients treated with BCG (7%), as well as immediate postoperative instillation of chemotherapy (<10%); in addition, there was no second-look transurethral resection (re-TUR) of the bladder was performed. The CUETO scoring model has been built based on a retrospective analysis of 1,062 patients underwent TUR of bladder tumor followed by 6-month BCG maintenance therapy. Nevertheless, the study was limited by the relatively old grading systems, lack of re-TUR or immediate intravesical instillation, and inadequacy for determining the time of recurrence.

Pan et al have developed a prognostic nomogram from the retrospective analysis of 1366 patients with NMIBC classified according to the 2004 World Health Organization WHO/International Society of Urologic Pathology grading system. Similarly, this study was limited by the retrospective nature, lack of the current recommendations of immediate intravesical instillation, and lack of studying other different prognostic factors . Ali-El-Dein et al have constructed a nomogram for recurrence and progression based on a retrospective analysis of more than 1000 patients from a single institution. Nevertheless, there was heterogeneity on the adjuvant regimens, in addition, re-TUR were not performed in all patients.

Recently, Cambier et al have published their nomograms and risk stratification systems based on a data from 1812 patients with intermediate risk and high risk NMIBC with adjuvant BCG maintenance therapy 1-3 years. Although this study presents the first prognostic factor analysis in NMIBC patients receiving the currently recommended 1-3 yr of maintenance BCG, it has several limitations. There was no repeat transurethral resection in high risk patients during the study period. In addition, there was no central pathology review, and there was no data on upper tract status at time of recurrence or progression.

Although all previously mentioned nomograms have demonstrated significant ability for detecting the outcome after transurethral resection of bladder tumor. Neither of these papers has included any other biological markers that have been proven to improve the predictive ability. Recently, special emphasis has been focused on the relation between smoking with recurrence and progression of NMIBC. It has been shown that smoking not only increases the risk of disease recurrence and progression, but also Current and heavy long-term smokers seem to be at the greatest risk for both end points. In addition, Ogihara et al have shown that a positive smoking history was an independent predictor for NMIBC recurrence and refraining from smoking for 15 years or more reduced the risk of tumor recurrence in former smokers with regardless of the intensity or duration of smoking.

Inflammation in the tumor microenvironment plays a crucial role in the proliferation and survival of malignant cells through enhanced angiogenesis, invasion, and metastasis. The underlying mechanisms include recruitment of T lymphocytes, chemokines, activated cytokines, secretion of CRP, and neutrophilia . In a recent meta-analysis, Masson-Lecomte et al have shown that among different inflammatory predictors, serum levels of C-reactive protein (CRP), Neutrophil to lymphocyte ratio (NLR), and urinary and serum interleukin levels were the most prognostic factors for bladder cancer prognosis. Furthermore, Kamat et al have shown that a cytokine panel had the potential for identifying patients at risk of tumor recurrence during BCG treatment. In addition, interleukin IL-2 have been shown to be the most prognostic biomarker for response to BCG therapy.

In a recent meta-analysis including 15,215 patients, Martin-Doyle et al have shown that the highest impact risk factor was depth of invasion into lamina propria. In addition, lymphovascular invasion, associated carcinoma in situ, tumor size > 3 cm, and older age were independent predictors for progression and cancer specific survival.

Currently, all publications investigating the outcome after treatment of NMIBC lack several factors including the re-staging TUR, maintenance BCG therapy, inclusion of other highly prognostic factors e.g. smoking, inflammatory biomarkers, depth of lamina invasion. Therefore, this protocol is constructed to combine all clinically affordable biomarkers into a prognostic model for predicting the outcome after NMIBC.

ELIGIBILITY:
Inclusion Criteria:

-Patient with NMIBC

Exclusion Criteria:

* Refuse to complete study requirements
* Contraindication to BCG therapy
* Muscle invasive disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible patient presented with NMIBC will be asked to participate in this study and will be provided with an informed consent form in line with Good Clinical Practise and the Declaration of Helsinki.
Sampling Method: Probability Sample
Enrollment: 761 (Estimated)
Dates: Start 2017-05-15 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Construct a new prognostic model for the prediction of recurrence and progression of NMIBC | 2 years
  Outcome Measure by counting and cmparing number of patients surviving for two year without tumor recurrence or progression to muscle invasive bladder cancer

SECONDARY OUTCOMES:
cancer-specific survival (CSS) after treatment of NMIBC | 5 years
  Outcome Measure by counting and comparing number of patients surviving for five year without tumor. Mortality cases will be counted if oncology is the cause of mortality
overall survival (OS) after treatment of NMIBC | 5 years
  Outcome Measure by conting and comparing number of patients surviving for five year without tumor. Mortality cases will be counted if the cause of mortality is other than oncology

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mosbah, MD, Study Chair — Urology and Nephrology Center
Locations (1):
- Urology and Nephrology Center, Mansora, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
meta-analyses by contact the Prof. Ahmed Mosbah MD (Study Chair)